CLINICAL TRIAL: NCT03504696
Title: Effectiveness, Safety and Use of Nivolumab Administered During the French Temporary Authorization for Use in Patients With Advanced (Unresectable or Metastatic) Melanoma: A Multicentric, Observational Study
Brief Title: Effectiveness, Safety and Use of Nivolumab Administered During the French Temporary Authorization for Use in Patients With Advanced Melanoma
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-555
Record Dates: First submitted 2018-02-22; First posted 2018-04-20 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Advanced Melanoma: RIC-Mel patients with advanced (unresectable or metastatic) melanoma treated with nivolumab in the context of nivolumab ATU program (occurred from 12-Sep-2014 to 31-Aug-2015)
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
This study will be conducted with the aim of estimating the effectiveness, safety, patterns of use of nivolumab, and characteristics of patients with unresectable or metastatic melanoma, treated with nivolumab monotherapy in the ATU setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in RIC-Mel Database:

  * Diagnosed with melanoma and cared for in the participating sites
  * Patients who have been given appropriate information about RIC-Mel Database aims and who have provided their written consent for data collection and processing before any data collection is carried out
* Patients included in French nivolumab ATU program

Exclusion Criteria:

• Patients included in RIC-Mel database having initiated nivolumab before 12-Sep-2014 or after 31-Aug-2015, or in the context of a clinical trial

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RIC-Mel patients with advanced (unresectable or metastatic) melanoma treated with nivolumab in the context of nivolumab ATU program (occurred from 12-Sep-2014 to 31-Aug-2015).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) at 1 year | at 1 year
  Overall survival (OS) for adult patients with advanced (unresectable or metastatic) melanoma treated with nivolumab in the ATU (Temporary Authorization for Use) program
Distribution of demographic characteristics of patients with advanced melanoma treated with nivolumab monotherapy in the ATU program | at baseline
  Distribution of demographic characteristics of patients with advanced melanoma treated with nivolumab monotherapy in the ATU program using descriptive statistics
Distribution of clinical characteristics in patients with advanced melanoma treated with nivolumab monotherapy | at baseline
  Clinical characteristics will be summarized using descriptive statistics.
Overall survival (OS) at 2 years | at 2 years
  Overall survival (OS) for adult patients with advanced (unresectable or metastatic) melanoma treated with nivolumab in the ATU (Temporary Authorization for Use) program

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year and 2 years
  (PFS) will be measured by the time since nivolumab initiation to either the first disease progression date or last known tumor assessment date, or death
Objective response rate (ORR) | 1 year and 2 years
  ORR is the proportion of patients with an objective response. Objective response is measured by the sum of partial responses plus complete responses as assessed by (RECIST 1.1) Response Evaluation Criteria In Solid Tumors
Progression-free survival (PFS) as assessed by RECIST 1.1 | at 1 year
  PFS measured by time since index date (initial treatment with nivolumab) to either the first disease progression date or last known tumor assessment date, or death due to any cause, whichever occurs first as assessed by RECIST 1.1
Distribution of treatment patterns | up to 2 years
  Details on Prior and Evolution of Current Treatment Patterns will be summarized using descriptive statistics.
Incidence of select Grade 3, 4, or 5 adverse events (AEs) | up to 2 years
  Select AEs include pulmonary, endocrine, gastrointestinal, hepatic, renal, cutaneous, and infusion reactions

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Nantes, France

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx